CLINICAL TRIAL: NCT00812188
Title: A Prospective, Open Label Trial of High Dose UVA-1, 3x/Week or Medium Dose UVA-1, 3x/Week vs. Fluocinonide 0.05% Cream Treatment of Morphea
Brief Title: Treatment Study Comparing Medium or High Dose Uva-1 Treatment 3x/Week Versus Fluocinonide 0.05% Cream in the Treatment of Morphea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Heidi Jacobe, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112004027
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2014-12

CONDITIONS: Symmetric Limited Morphea
Keywords: Morphea; Plaque morphea; Localized Scleroderma
MeSH Terms: conditions — Scleroderma, Localized

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medium Dose UVA-1 (Active Comparator): Medium dose (60 J/cm2) UVA-1 3x/week for 12 weeks to one morphea plaque and fluocinonide 0.05% cream to another morphea plaque twice daily for twelve weeks.
  Interventions: Other: Medium Dose UVA-1
- High Dose UVA-1 (Active Comparator): High dose UVA-1 treatment 3x/week for 12 weeks to one morphea plaque and fluocinonide 0.05% cream twice daily for 12 weeks to another morphea plaque.
  Interventions: Other: High Dose UVA-1

INTERVENTIONS:
Other: Medium Dose UVA-1 — UVA-1 phototherapy treatment (60 J/cm2) three times per week for 12 weeks.
  Arms: Medium Dose UVA-1
Other: High Dose UVA-1 — High dose (120 J/cm2)UVA-1 phototherapy three times per week for 12 weeks.
  Arms: High Dose UVA-1

SUMMARY:
Compare UVA-1 phototherapy treatment to topical steroid treatment in subjects with morphea.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older.
* Symmetric limited morphea.

Exclusion Criteria:

* Known sensitivity to fluocinonide 0.05% cream.
* Clinical evidence of superinfected skin.
* Immunocompromised state (including previously documented HIV).
* Generalized Scleroderma.
* Previous history of skin cancer.
* Non-English speaking subjects.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of UVA-1 treatment vs. topical steroid. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Jacobe, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas - Department of Dermatology Clinical Trials, Dallas, Texas, United States